CLINICAL TRIAL: NCT03652428
Title: Phase I Study of Concurrent Nab-Paclitaxel + Gemcitabine With Hypofractionated, Ablative Proton Therapy for Locally Advanced Pancreatic Cancer
Brief Title: Phase I Nab-Paclitaxel Plus Gemcitabine With Proton Therapy for Locally Advanced Pancreatic Cancer (LAPC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00081403
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: LAPC; Nab-paclitaxel +Gemcitabine; Proton Therapy
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pancreatic Proton Therapy With Concurrent Gem + Nab-paclitaxel (Other): Part I:
  Gemcitabine + nab-paclitaxel:
  • Administered per institutional standard every 7 days for 3 weeks
  Part II:
  Hypofractionated ablative pancreatic proton radiation therapy 67.5 Gy fractions once per day Monday - Friday for 3 weeks, for a total of 15 fractions.
  Part III:
  Surgery, if resectable, then adjuvant chemo per discretion of MD or no further therapy
  OR
  Chemo per discretion of MD if not resectable
  Interventions: Drug: Gemcitabine; Radiation: Hypofractionated Ablative Proton Therapy

INTERVENTIONS:
Drug: Gemcitabine — see arm description
  Other Names: Nab-Paclitaxel
Radiation: Hypofractionated Ablative Proton Therapy — see arm description

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of the chemotherapy drugs nab-paclitaxel and gemcitabine when combined with hypofractionated ablative proton therapy for the treatment of locally advanced pancreatic cancer. You will receive proton therapy once a day (Monday - Friday) for 3 weeks. Participants will also receive chemotherapy on each Monday of those three weeks.

DETAILED DESCRIPTION:
The investigators propose a phase I trial to determine the maximum tolerable dose (MTD) and the recommended dose for phase II (RP2D) of concurrent nab-paclitaxel + gemcitabine in combination with ablative IMPT delivered as a fixed dose of 67.5 Gy in 15 fractions daily fractions with 5 fractions per week. In contrast to prior pancreatic cancer studies of chemoradiotherapy which utilized photon RT to treat gross disease and elective lymph nodes (1,2) the proposed study is hypothesized to reduce toxicity risk by limiting highly conformal IMPT to the gross tumor volume. Furthermore, to increase the margin of safety in a manner similar to published data from MDACC (3), the high dose region will be limited to areas at least 5 mm from nearby GI structures (duodenum, small bowel, stomach, etc.). Regions within this area will be treated only to 37.5 Gy in 15 fractions. This dose limitation is also important given that paclitaxel, in addition to increasing systemic efficacy, is a known radiosensitizer (1).

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreas.
2. Nonmetastatic pancreatic cancer. Metastatic disease includes spread to distant (non-regional) lymph nodes, organs, peritoneum and ascites.
3. Unequivocal radiographic findings contraindicating resection including, but not limited to, solid tumor contact with any of the following: 1) the SMA >180º; 2) the celiac axis >180º; 3) the first jejunal superior mesenteric artery (SMA) branch; 4) unreconstructible superior mesenteric vein (SMV)/portal vein due to tumor involvement or occclusion; 5) the most proximal draining jejunal branch into the SMV.
4. ECOG Performance Status 0 or 1.
5. Absolute neutrophil count ≥1,000/mm3
6. Platelet count ≥100,000/mm3
7. Creatinine ≤1.5 × upper limit of normal
8. Calculated creatinine clearance >45 mL/min
9. Total bilirubin ≤2 mg/dL

Exclusion Criteria:

1. Patients with resectable or borderline resectable pancreatic cancer are ineligible.
2. No prior definitive resection of pancreatic cancer.
3. No prior radiation therapy to the abdomen that would overlap fields required in this study. Prior radiotherapy for other disease is allowed.
4. No prior chemotherapy except for FOLFIRINOX, Gem-Abrax, or Gem-Cap. A patient may be registered for the trial while undergoing chemotherapy.
5. Any grade 4 toxicity prior to start of chemoradiotherapy that may be due to induction chemotherapy.
6. Greater than 2 dose reductions during induction chemotherapy.
7. Chronic concomitant treatment with strong inhibitors of CYP3A4. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to the start of study treatment. Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment.
8. Baseline Grade ≥ 2 neuropathy. Known Gilbert's disease or known homozygosity for UGAT1A1*28 polymorphism.
9. Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry if they are in childbearing years/premenopausal.
10. Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with gemcitabine and nab-paclitaxel.
11. Non-compliance with induction chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Gemcitabine and nab-Paclitaxel in LAPC patients receiving proton therapy | Patients will be followed for 12 months after registration or until death, whichever occurs first.
  Maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy for the treatment of locally advanced pancreatic cancer.

SECONDARY OUTCOMES:
Primary Tumor Response in LAPC patients receiving proton therapy with concurrent Gemcitabine and nab-Paclitaxel | Patients will be followed for 12 months after registration or until death, whichever occurs first.
  Primary tumor response in patients receiving with LAPC receiving preoperative concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy evaluated by CT or MRI
Survival status (disease-free-survival vs. overall survival) | Patients will be followed for 12 months after registration or until death, whichever occurs first.
  Time to recurrence and site of recurrence in patients with LAPC receiving preoperative concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy (RECIST)
Median Overall Survival of Patients | Patients will be followed for 12 months after registration or until death, whichever occurs first.
  Median overall survival of patients with LAPC receiving preoperative concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy
R0 Resection | Patients will be followed for 12 months after registration or until death, whichever occurs first.
  R0 resection rates in patients with LAPC receiving preoperative concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy
Number of adverse events/toxicites reported during and following treatment of concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy | Patients will be followed for 12 months after registration or until death, whichever occurs first.
  Number of toxicities participants reported by participants during and following treatment of concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy (NIH CTCAE v 4)
Quality of life through and after treatment | Patients will be followed for 12 months after registration or until death, whichever occurs first.
  Patient reported quality of life impact from receiving preoperative concurrent nab-paclitaxel + gemcitabine combined with hypofractionated ablative proton therapy using the FACT-Hep questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jason Molitoris, MD, Principal Investigator — University of Maryland/Maryland Proton Treatment Center
Locations (2):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Maryland Medical Center/Maryland Proton Treatment Center, Baltimore, Maryland

REFERENCES:
- [Background] Rich T, Harris J, Abrams R, Erickson B, Doherty M, Paradelo J, Small W Jr, Safran H, Wanebo HJ. Phase II study of external irradiation and weekly paclitaxel for nonmetastatic, unresectable pancreatic cancer: RTOG-98-12. Am J Clin Oncol. 2004 Feb;27(1):51-6. doi: 10.1097/01.coc.0000046300.88847.bf. PMID 14758134
- [Background] Crane CH, Janjan NA, Evans DB, Wolff RA, Ballo MT, Milas L, Mason K, Charnsangavej C, Pisters PW, Lee JE, Lenzi R, Vauthey JN, Wong A, Phan T, Nguyen Q, Abbruzzese JL. Toxicity and efficacy of concurrent gemcitabine and radiotherapy for locally advanced pancreatic cancer. Int J Pancreatol. 2001;29(1):9-18. doi: 10.1385/IJGC:29:1:09. PMID 11560155
- [Background] Krishnan S, Chadha AS, Suh Y, Chen HC, Rao A, Das P, Minsky BD, Mahmood U, Delclos ME, Sawakuchi GO, Beddar S, Katz MH, Fleming JB, Javle MM, Varadhachary GR, Wolff RA, Crane CH. Focal Radiation Therapy Dose Escalation Improves Overall Survival in Locally Advanced Pancreatic Cancer Patients Receiving Induction Chemotherapy and Consolidative Chemoradiation. Int J Radiat Oncol Biol Phys. 2016 Mar 15;94(4):755-65. doi: 10.1016/j.ijrobp.2015.12.003. Epub 2015 Dec 11. PMID 26972648